CLINICAL TRIAL: NCT02221128
Title: A Post Market Surveillance Study Evaluating the Safety and Effectiveness of PerClot to Control Mild Bleeding in Subjects Undergoing Endoscopic Sinus Surgery
Brief Title: PerClot to Control Bleeding in Endoscopic Sinus Surgery
Status: Completed | Type: Observational
Sponsor: CryoLife Europa (Industry)
Collaborators: CryoLife, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: PCT1402.001M(06/14)
Record Dates: First submitted 2014-07-03; First posted 2014-08-20 (Estimated); Last update posted 2014-10-03 (Estimated); Status verified 2014-07

CONDITIONS: Sinusitis
MeSH Terms: conditions — Sinusitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
A prospective, single centre, single arm study designed to collect clinical data on PerClot when used in subjects undergoing endoscopic sinus surgery.

ELIGIBILITY:
Inclusion Criteria:

* Subjects having Endoscopic Sinus Surgery
* Subjects who will have PerClot used as a haemostatic agent
* Subjects willing and able to give consent
* Subjects over 18 years old

Exclusion Criteria:

* Subjects unable or unwilling to give consent for their data to be collected

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults undergoing Endoscopic Sinus Surgery
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2014-07; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Number of subjects who achieve of haemostasis after the application of PerClot | intraoperatively

SECONDARY OUTCOMES:
Number of subjects who require the use of alternative methods to achieve haemostasis after the application of PerClot | intraoperatively

CONTACTS AND LOCATIONS:
Overall Officials: David Roberts, Principal Investigator — Guy's and St Thomas' NHS Foundation Trust
Locations (1):
- Guys and St Thomas NHS Trust, London, United Kingdom